CLINICAL TRIAL: NCT00676481
Title: Rapid HIV Testing for Emergency Department Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: K23 A1060363; K23 A1060363; U65/CCU124504
Record Dates: First submitted 2008-05-09; First posted 2008-05-13 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2008-05

CONDITIONS: HIV Infections
Keywords: Patient Education; Emergency Medicine; HIV Prevention; HIV Seronegativity
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Phase III participants who are educated about risk of HIV infection before receiving a rapid HIV test
  Interventions: Behavioral: HIV risk education
- 2 (No Intervention): Phase III participants who are not educated about risk of HIV infection before receiving a rapid HIV test

INTERVENTIONS:
Behavioral: HIV risk education — Education for Phase III participants about potential risk of HIV infection before being asked to take a rapid HIV test in the ED
  Arms: 1

SUMMARY:
The purpose of this study is to test data collection options in emergency departments (EDs) and to enhance ED patient awareness of the risk of HIV infection.

DETAILED DESCRIPTION:
Rapid HIV testing is a new technology that speeds receipt of HIV test results. Its use in EDs has been demonstrated, but patient acceptance of rapid testing in the ED has not been optimal. It is likely that the low acceptance is partially due to ED patients not realizing the risk of acquiring an HIV infection or the importance of knowing their HIV status. The purpose of this study is to test data collection options in EDs and to enhance ED patient awareness of the risk for HIV infection.

This three phase study will take place at the Rhode Island Hospital Emergency Department. Each participant will be followed for the duration of their ED visit.

In Phase I, the proportion of participants who are willing to undergo rapid HIV testing in the ED will be measured. Additionally, the HIV testing history of these participants, their reasons for undergoing testing or for never having been tested for HIV, and factors associated with acceptance or decline of testing and history of HIV testing will be determined. An educational video will be developed and used to investigate its effectiveness in convincing participants to have the rapid HIV test. All participants agreeing to undergo a rapid HIV test will receive a survey to complete.

In Phase II, a questionnaire and feedback tool to make participants aware of their risk for an HIV infection through injection drug use and sex will be developed and investigated.

In Phase III, the questionnaire and feedback tool developed in Phase II will be used to determine whether or not making participants aware of their risk for an HIV infection increases their acceptance of being tested for HIV in the ED. Participants in Arm 1 will receive the questionnaire and feedback tool while participants in Arm 2 will not.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Subcritical illness or injury

Exclusion Criteria:

* Critical illness or injury
* Mental or physical disability
* Known HIV infection
* Participation in an HIV vaccine study
* Prison inmate
* Acute psychiatric illness that, in the opinion of the investigator, would prevent the participant from completing the study

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 570 (Actual)
Dates: Start 2004-07; Primary Completion 2009-03 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Willingness of participant to have HIV testing | Throughout study

SECONDARY OUTCOMES:
Participant comprehension of rapid HIV pre-test information | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Roland C Merchant, MD, MPH, ScD, Principal Investigator — Rhode Island Hospital/Warren Alpert Medical School
Locations (1):
- Rhode Island Hospital Emergency Department, Providence, Rhode Island, United States